CLINICAL TRIAL: NCT06598969
Title: Phase II Study of TMLI Administered in Combination With a Myeloablative Regimen (Cyclophosphamide + Etoposide) for Allogeneic Hematopoietic Stem Cell Transplantation in Patients With High-risk Myelodysplastic Syndrome or Acute Myeloid Leukemia
Brief Title: TMLI Plus Chemotherapy in High Risk Myelodysplastic Syndrome or Acute Myeloid Leukemia
Acronym: TMLI-MA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TMLI-MA
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Myelodysplastic Syndromes; Myeloid Leukemia, Acute
Keywords: High-Risk myelodysplastic syndrome; Acute myeloid leukemia; Total narrow and lymphoid irradiation
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Lymphatic Irradiation

STUDY DESIGN:
Intervention Model Description: To evaluate the antileukemic activity and safety/tolerability of the TMLI/cyclophosphamide and etoposide conditioning regimen followed by allogeneic hematopoietic stem cell transplantation in patients with high-risk myelodysplastic syndrome or acute myeloid leukemia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): This trial is designed to evaluate the antileukemic activity of an Total bone marrow and lymphoid irradiation/cyclophosphamide/etoposide conditioning regimen for allogeneic hematopoietic stem cell transplantation, in patients with high-risk myelodysplastic syndromes and acute myeloid leukemia, as assessed by 2-year progression-free survival. The first 6-18 patients enrolled/treated in this study will be part of a safety sub-analysis, so patients will be assigned to the dose level that is currently open once they are verified to be eligible; up to three dose levels can be studied.
  Interventions: Drug: Total bone marrow and lymphoid irradiation/cyclophosphamide/etoposide

INTERVENTIONS:
Drug: Total bone marrow and lymphoid irradiation/cyclophosphamide/etoposide — Evaluate the antileukemic activity of an total bone marrow and lymphoid irradiation/cyclophosphamide/etoposide conditioning regimen for allogeneic hematopoietic stem cell transplantation

SUMMARY:
Single-arm, single-center phase II trial to evaluate the antileukemic activity and safety/tolerability of TMLI/cyclophosphamide and etoposide conditioning regimen followed by allogeneic hematopoietic stem cell transplantation in patients with high-risk myelodysplastic syndrome or acute myeloid leukemia.

DETAILED DESCRIPTION:
The aim of this study is the evaluation of the antitumor activity of the conditioning regimen with TMLI, cyclophosphamide and etoposide followed by allogeneic hematopoietic stem cell transplantation by means of the progression-free survival at 2 years after a safety-lead phase.

The determination of the complete remission rate at day 30 post-transplant, the estimation of overall survival, the cumulative incidence of recurrence/progression, and non-relapse mortality at 100 days, 1 year, and 2 years, the Minima Residual Disease monitoring at 30, 90, 180, 270 days and 1 year, 1 year and a half and 2 years post-transplant, and the assessment early and late toxicities/complications by organ and severity, as well as dose/dose-volume toxicity characterization across organs, including acute/chronic graft-versus-host disease, infection, and long-term complications are included as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* The participant has the ability and willingness to sign the informed consent document
* Age ≥18 to ≤50 years.
* Karnofsky's performance status should be ≥70%.
* Patients with myelodysplastic syndrome/acute myeloid leukemia or acute myeloid leukemia with relapsed/refractory active disease, or in complete remission or morphologic leukemia-free state with evidence of measurable residual disease as assessed by multiparameter flow cytometry (≥ 0,1%) or next-generation sequencing
* All candidates for this study must have an Human leukocyte antigens (A, B, C, DR) identical siblings who are willing to donate bone marrow or peripheral blood hematopoietic progenitors or an 8/8 matched unrelated donor. A single allele mismatch in A, B, C or DR beta chain 1 shall be allowed
* Total bilirubin ≤ 1.5 x upper limit of normal or 3 x upper limit of normal for Gilbert's disease.
* serum glutamate oxaloacetate transaminase & serum glutamate pyruvate transaminaseT ≤ 5 x upper limit of normal.
* Serum creatinine ≤ 1.3 mg/dL or creatinine clearance measured ≥ 80 mL/min for 24 hours of urine collection
* Women of childbearing age only: Negative urine or serum pregnancy test
* Pulmonary function tests: forced expiratory volume in one second and Carbon Monoxide Diffusion Capacity (adjusted for Hb) ≥ 50% from expected normal value
* Patients should undergo cardiac evaluation with an electrocardiogram showing no ischemic changes or clinically relevant arrhythmia, and a ≥50% ejection fraction established by Multi-Gated Acquisition Scan or echocardiogram
* Men and women of childbearing potential agree to use appropriate contraceptives (hormonal or barrier contraception or abstinence) prior to study entry and for six months following the duration of study participation
* The time elapsed since the end of the last induction or reinduction cycle must be greater than or equal to 14 days

Exclusion Criteria:

* Patients who have received a previous autologous (within the last year) or allogeneic transplant (at any time) are excluded
* Previous radiation therapy, which would preclude the use of total bone marrow and lymphoid irradiation
* Plans during the trial to receive any other investigational (non-trial-related) agents
* Uncontrolled disease, including ongoing or active infection
* History of allergic reactions attributed to compounds of chemical or biological composition similar to cyclophosphamide or etoposide
* Patients with other active malignancies are not eligible for this study, other than the malignancies discussed
* Patients with a psychological or medical condition that the patient's physician deems unacceptable to proceed with allogeneic hematopoietic stem cell transplantation
* Women who plan to become pregnant or breastfeed during the trial
* Patients who do not agree to practice effective forms of contraception
* Subjects who, in the opinion of the investigator, may not be able to meet the safety control requirements of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From the start of therapy to 2 years after post-transplant
  Time from the start of treatment to the date of death, disease relapse/progression, or date of last follow-up.

SECONDARY OUTCOMES:
Overall survival | From the start of therapy to 2 years after post-transplant
  Quantification of time of patients who are still alive
Cumulative incidence of recurrence/progression | From the start of therapy to 2 years after post-transplant
  The event is relapse/progression either extramedullary or at bone marrow
Complete remission rate | From the day of infusion to the day 30 post-transplant
  The event is whether or not the patient has a documented complete remission
Non-relapse mortality | From the start of therapy until 2 years after post-transplant
  Number of deaths from causes other than relapse or progression
Measurable residual disease | At 30, 90, 180 days and 1 year, 1.5 year and 2 years post-transplant
  Measurable residual disease monitoring assessed by multiparameter flow cytometry
Incidence of infection | 2 years after post-transplant
  Describe the infections.
Adverse Events | 2 years after post-transplant
  Describe the adverse event
Acute graft-versus-host disease grades 2-4 and 3-4 | 100 days post-transplant
  This point is classified according to the consensus MAGIC classification
Chronic graft-versus-host disease | 2 years after post-transplant
  Describe the chronic graft-versus-host disease according to the National Institutes of Health Stroke Scale consensus staging.

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio Pérez Simón, MD-PhD, Principal Investigator — Fundación para la Gestión de la Investigación en Salud de Sevilla
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Spain

IPD SHARING:
Plan to Share IPD: No